CLINICAL TRIAL: NCT02562885
Title: Effect of Closed-loop Auditory Stimulation on Spike Waves During Slow Wave Sleep, an Open Label Pilot Study
Brief Title: Effect of Auditory Stimulation on Spike Waves in Sleep
Acronym: ECLASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SW2015
Record Dates: First submitted 2015-09-21; First posted 2015-09-29 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2016-12

CONDITIONS: Epilepsy; Sleep
Keywords: Benign epilepsy with centro-temporal spikes; Continuous spike waves in slow wave sleep; Electroencephalography; Sleep, slow wave
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acoustic pulses (Experimental): During NREM sleep:
  1. 15 minutes without acoustic pulses
  2. 15 minutes with acoustic pulses
  3. 15 minutes without acoustic pulses
  Two different protocols are applied:
  (A) tone application at the "Down-phase" of sleep slow wave (SSW) (B) tone application at the "Up-phase" of SSW.
  Participants with Rolandic epilepsy/BECTS or generalized spike waves: Protocol A and B alternatingly.
  Participants with ESES/CSWS: only Protocol A.
  Interventions: Device: Acoustic pulses

INTERVENTIONS:
Device: Acoustic pulses — Acoustic pulses applied during NREM sleep slow waves "Up-phase" or "Down-phase". The acoustic stimulus will be delivered by speakers with a volume of about 50 dB.

SUMMARY:
Background: Close relationship exists between sleep slow wave (SSW) and the generation of spike wave in NREM-sleep. SSW are cortically generated oscillations alternating between excitatory depolarization ("Up-phase" of the SSW) and inhibitory hyperpolarization ("Down-phase" of the SSW). It has been shown experimentally that with increasing synchrony of slow neuronal oscillations SSW turn into spike waves. Acoustic pulses applied in correspondence to the SSW "Up-phase" enhance the amplitude of the subsequent SSW. Conversely, tones delivered at the SSW "Downphase" have a disruptive effect on the following SSW.

Participants: Patients with epilepsy and spike waves in NREM-sleep.

Objective: Modification of spike wave frequency, amplitude and spreading during NREM sleep by acoustic pulses applied at the "Up-" or "Down-phase" of SSW.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Rolandic epilepsy/BECTS
* Participants with ESES/CSWS
* Participants with generalized spike waves in sleep
* EEG within 6 months before study night consistent with the diagnosis

Exclusion Criteria:

* Clinically significant concomitant acute or chronic disease
* Seizure frequency >1/week, history of convulsive status epilepticus or seizures provoked by sleep deprivation
* Severe sleep problems
* Treatment with corticosteroids, immunosuppressive or vagus nerve stimulation

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Spike wave index | Change baseline (without) and with acoustic pulses in the same NREM period: 45 minutes
  Change of spike wave index during acoustic pulses applied at the "Up-" or "Down-phase" of sleep slow waves. Spike wave index given in percent and calculated by number of seconds within 10 second windows with spike waves over the whole 15 minutes of the block design part.

SECONDARY OUTCOMES:
Spike wave amplitude | Change baseline (without) and with acoustic pulses in the same NREM period: 45 minutes
  Change of spike wave amplitude (in microvolts) during acoustic pulses applied at the "Up-" or "Down-phase" of sleep slow waves. Amplitudes of maximum spike will be analyzed in 10 seconds periods of the first and the last 100 seconds of every part of the block design. EEG source derivation will be used for the analysis. The mean of the 3 highest amplitudes of each 10 seconds period will be determined and the mean of the 10 periods will presented in mean and SD.
Spike wave spreading | Change baseline (without) and with acoustic pulses in the same NREM period: 45 minutes
  Change of spike wave spreading during acoustic pulses applied at the "Up-" or "Down-phase" of sleep slow waves. Spreading will be analyzed in 10 seconds periods of the first and the last 100 seconds of every part of the block design. EEG source derivation will be used for the analysis. Maximum spike wave spreading (number of electrodes involved) visible in 3 spike waves of each 10 second period will be determined and the mean of the 10 periods will presented in mean and SD.
Spike wave index in the NREM (2) period following the NREM (1) period with acoustic pulses | Change baseline (NREM 1) and NREM 2: expected average of 1 hour
  Change of spike wave index in the NREM period following the NREM period with acoustic pulses applied at the "Up-" or "Down-phase" of sleep slow waves. Over the first 15 minutes of the following NREM period: Spike wave index given in percent and calculated by number of seconds within 10 second windows with spike waves .
Spike wave amplitude in the NREM (2) period following the NREM (1) period with acoustic pulses | Change baseline (NREM 1) and NREM 2: expected average of 1 hour
  Change of spike wave amplitude (in microvolts) in the NREM period following the NREM period with acoustic pulses applied at the "Up-" or "Down-phase" of sleep slow waves. Amplitudes of maximum spike will be analyzed in 10 seconds periods of the first and the last 100 seconds of the following NREM period. EEG source derivation will be used for the analysis. The mean of the 3 highest amplitudes of each 10 seconds period will be determined and the mean of the 10 periods will presented in mean and SD.
Spike wave spreading in the NREM (2) period following the NREM (1) period with acoustic pulses | Change baseline (NREM 1) and NREM 2: expected average of 1 hour
  Change of spike wave spreading in the NREM period following the NREM period with acoustic pulses applied at the "Up-" or "Down-phase" of sleep slow waves. Spreading will be analyzed in 10 seconds periods of the first and the last 100 seconds of the following NREM period. EEG source derivation will be used for the analysis. Maximum spike wave spreading (number of electrodes involved) visible in 3 spike waves of each 10 second period will be determined and the mean of the 10 periods will presented in mean and SD.

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Schmitt, MD, Principal Investigator — Div. of Clinical Neurophysiology/Epilepsy, University Children's Hospital, Steinwiesstrasse 75, CH-8032 Zurich
Locations (1):
- Div. of Clinical Neurophysiology/Epilepsy, University Children's Hospital Zurich, Zurich, Switzerland